CLINICAL TRIAL: NCT04899661
Title: Long-term Special Drug Use Investigation of Molidustat for Patients With Renal Anemia
Brief Title: A Study to Learn More About the Long-term Safety and Effectiveness of Molidustat as a Treatment for Japanese Men and Women With Renal Anemia
Status: Active, not recruiting | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 21319
Record Dates: First submitted 2021-05-20; First posted 2021-05-24 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Renal Anemia
MeSH Terms: interventions — molidustat

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Molidustat: Participants diagnosed with renal anemia treated with Molidustat at the discretion of investigators
  Interventions: Drug: Molidustat (Musredo, BAY85-3934)

INTERVENTIONS:
Drug: Molidustat (Musredo, BAY85-3934) — Tablets, administered orally at the discretion of investigators

SUMMARY:
In this study, the researchers want to learn more about the safety and effectiveness of Molidustat in Japanese men and women who have renal anemia, a condition in which the kidneys do not make enough of a hormone that helps the body make new red blood cells.

In previous clinical trials with a small number of participants, several important adverse events were observed. The researchers in this study want to know how many patients also have these adverse events under the real world, and if the number of the red blood cells will be increased after the treatment of Molidustat.

The researchers will collect the participants' health information from their medical records and their regular check-ups for up to 2 years. The data from this study will be submitted to the health authority in Japan in accordance with the local regulation.

ELIGIBILITY:
Inclusion Criteria:

* Female or male participants with a diagnosis of renal anemia
* Decision to initiate treatment with Molidustat was made as per investigator's routine treatment practice
* Molidustat naïve participants (with including the participants treated within three months before the contracted date at each site)
* Signed informed consent

Exclusion Criteria:

- Contra-indications according to the local marketing authorization

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with a diagnosis of renal anemia and have been prescribed Molidustat in accordance with the product label
Sampling Method: Non-Probability Sample
Enrollment: 1081 (Actual)
Dates: Start 2021-08-06 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of safety events | Up to approximately 24 months
  Adverse Events/Adverse Drug Reactions including thromboembolism, hypertension, malignant tumor retinal hemorrhage, Major Adverse Cardiovascular Events (MACE) without thromboembolism, Interstitial lung disease (ILD) and Progression of Autosomal Dominant Polycystic Kidney Disease (ADPKD) in renal anemia patients

SECONDARY OUTCOMES:
Incidence of safety events in dialysis and non-dialysis participants | Up to approximately 24 months
  Adverse Events/Adverse Drug Reactions including thromboembolism, hypertension, malignant tumor retinal hemorrhage, Major Adverse Cardiovascular Events (MACE) without thromboembolism, Interstitial lung disease(ILD) and Progression of Autosomal Dominant Polycystic Kidney Disease (ADPKD) in renal anemia patients
Incidence of safety events (important identified risk and important potential risk) by patient background | Up to approximately 24 months
  Important identified risk: "Thromboembolism" and "Hypertension"
  Important potential risk:
  "Malignant tumor", "Retinal hemorrhage", "Major Adverse Cardiovascular Events (MACE) without thromboembolism", "Interstitial lung disease(ILD)" and "Progression of Autosomal Dominant Polycystic Kidney Disease (ADPKD)"
Absolute changes of Hemoglobin (Hb) levels from the baseline | Up to approximately 24 months
Percentage changes of Hemoglobin (Hb) levels from the baseline | Up to approximately 24 months
Absolute changes of Hb levels from baseline in sub-group analysis | Up to approximately 24 months
  By patient background
Percentage changes of Hb levels from baseline in sub-group analysis | Up to approximately 24 months
  By patient background
Time course of Hb levels from the baseline | Up to approximately 24 months
Proportion of participants with Hb level within target range | Up to approximately 24 months

CONTACTS AND LOCATIONS:
Locations (1):
- Many facilities, Multiple Locations, Japan

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014. Interested researchers can use www.clinicalstudydatarequest.com to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the Study sponsors section of the portal.